CLINICAL TRIAL: NCT02418494
Title: Development of a Health-Related Symptom Index for Persons Diagnosed With and Either Treated or Monitored for Anal High-Grade Squamous Intraepithelial Lesions (HSIL)
Brief Title: Health-Related Symptom Questionnaires in Measuring Quality of Life in HIV-Infected Participants Treated or Monitored for Anal Lesions
Status: Completed | Type: Observational
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Memorial Sloan Kettering Cancer Center (Other); Northwestern University (Other); The Emmes Company, LLC (Industry); University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: AMC-A02; NCI-2015-00160 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC Protocol #A02 (Other: AIDS Malignancy Clinical Trials Consortium); AMC-A02 (Other: AIDS Malignancy Clinical Trials Consortium); AMC-A02 (Other: CTEP); U01CA121947 (NIH)
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-02

CONDITIONS: High Grade Anal Canal Squamous Intraepithelial Neoplasia; HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (ANCHOR HRQoL interview, cognitive interview): Participants complete the ANCHOR HSIL HRQoL interview over 45-60 minutes, comparing the list of symptoms, concerns, or HRQOL impacts related to HSIL diagnosis and treatment. Some patients also undergo a cognitive interview for up to 3 sessions.
  Interventions: Other: Concept Elicitation; Other: Comprehension Assessment

INTERVENTIONS:
Other: Concept Elicitation — Complete cognitive interview to elicit relevant HSIL symptoms, compare to study index of symptoms, and rank symptoms in relation to effect on health-related quality of life
  Other Names: Cognitive Interview
Other: Comprehension Assessment — Comprehension assessment of draft quality of life assessment
  Other Names: Cognitive Interview

SUMMARY:
This research trial studies health-related symptom questionnaires in measuring quality of life in human immunodeficiency virus (HIV)-infected participants treated with or monitored for anal lesions. Collecting information and symptoms from patients diagnosed with anal lesions may help reduce the risk of anal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop an Anal Cancer/HSIL Outcomes Research Study (ANCHOR) high-grade squamous intraepithelial lesion (HSIL) health-related quality of life (HRQoL) Index (HQI) using state-of-the-art measure development methodology that captures the most important HRQoL symptoms and concerns of those persons diagnosed with anal HSIL and either treated or untreated for anal HSIL.

OUTLINE:

Participants complete the ANCHOR HSIL HRQoL interview over 45-60 minutes, comparing the list of symptoms, concerns, or HRQOL impacts related to HSIL diagnosis and treatment. Some patients also complete a cognitive interview for up to 3 sessions.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Biopsy-proven anal HSIL within the prior six months
* Life expectancy of greater than 5 years

Exclusion Criteria:

* History of anal cancer
* Inability to understand a written consent form

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with HSIL within the prior 6 months enrolled at Weill Cornell Medical College/New York Presbyterian Hospital, Montefiore Medical Center, and Laser Surgery Care Center
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Development of an HQI using state-of-the-art measure development methodology that captures the most important HRQoL symptoms and concerns of those persons diagnosed with anal HSIL and either treated or untreated for anal HSIL. | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jack Burkhalter, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (6):
- United States (6):
  - University of California at San Francisco - Comprehensive Cancer Center, San Francisco, California
  - Anal Dysplasia Clinic, Chicago, Illinois
  - Cornell Clinical Trials Unit, New York, New York
  - Laser Surgery Care, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York